CLINICAL TRIAL: NCT05511077
Title: Biomarkers of Oat Product Intake: The BiOAT Marker Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chalmers University of Technology (Other)
Collaborators: Oatly Group Inc (Unknown)
Responsible Party: Principal Investigator, Rikard Landberg, Professor, Chalmers University of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ChalmersU
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Healthy
MeSH Terms: interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liquid oat product (Other)
  Interventions: Other: Diet
- Solid oat product (Other)
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Intervention products consist of two different oat products, one solid and one liquid. The content of oat in the products differs.

SUMMARY:
The aim of this project is to evaluate avenanthramides and avenacosides and their metabolites as specific biomarkers of oat product intake in humans. Biomarkers will be evaluated after i) a single dose through a single meal based on a solid and a liquid oat-based product (pharmacokinetic study) ii) week-long consumption at three different intake levels (dose-response). The study will be carried out as a two-way cross-over design with two different oat products, liquid or solid, where each product is provided 3 times per day during 5 days per product. A wash-out period of 8 days where participants consume their habitual diet is implemented. The first day of study meal intervention includes postprandial measurements during 8 hours.

ELIGIBILITY:
Inclusion Criteria:

* Females and males
* Age 18-80 years
* Body mass index (BMI) 18.5-30 kg/m2
* Fasting glucose ≤ 6.1 mmol/l
* Low density lipoprotein (LDL) Cholesterol ≤ 5.30 mmol/L
* Triglycerides ≤ 2.60 mmol/L
* Signed informed consent

Exclusion Criteria:

* Food allergies or intolerances preventing consumption of any products included in the study.
* Unable to sufficiently understand written and spoken Swedish to provide written consent and understand information and instructions from the study personal.
* Pregnant, lactating or planning a pregnancy during the study period.
* Antibiotic use for the last 3 months.
* Blood donation or participation in a clinical study with blood sampling within 30 days prior to screening visit and throughout the study.
* History of stomach or gastrointestinal conditions (Inflammatory bowel disease, Crohn's disease, malabsorption, colostomy, bowel resection, gastric bypass surgery etc.)
* Previous major gastrointestinal surgery
* Have type I diabetes
* Thyroid disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of avenanthramides and avenacosides and their metabolites. | 24 hours
  Difference in the plasma concentrations of diet specific biomarkers comparing before (baseline) and after intervention meal (average plasma concentration over a 24 h period).
Plasma concentration-time profile over 24h (AUCs) of avenanthramides and avenacosides and their metabolites. | 24 hours
  Differences in plasma AUCs between the intake levels for each biomarker candidate.
Urine concentrations of avenanthramides and avenacosides and their metabolites | 8 hours
  Difference in the plasma concentrations of diet specific biomarkers comparing before (baseline) and after intervention meal (average urine concentration over a 8 h period).

SECONDARY OUTCOMES:
Gut microbiome | 5 days
  Fecal samples will analyzed for composition of the gut microbiome, baseline compared with after 5 days of intervention products.
Plasma metabolites | 5 days
  Untargeted metabolomics will be performed using established methods for plasma. Analyzed exploratorily using untargeted metabolomics to find potential biomarker panels that reflect oats product intake. Baseline compared with after intervention products.
Urine metabolites | 24 hours
  Untargeted metabolomics will be performed using established methods for urine. Analyzed exploratorily using untargeted metabolomics to find potential biomarker panels that reflect oats product intake.
Blood concentrations of avenanthramides and avenacosides and their metabolites | 8 hours
  Evaluate new simple sampling techniques using dried blood spots.

CONTACTS AND LOCATIONS:
Overall Officials: Rikard Landberg, Dr, Principal Investigator — Chalmers University of Technology
Locations (1):
- University of Gothenburg, Department of Food and Nutrition and Sport Science, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Armeni M, Cardilin T, Fristedt R, Karlsson T, Jenkins CO, Nordin E, Qin P, Jirstrand M, Kristiansen K, Savolainen O, Landberg R. Avenanthramides and avenacosides as biomarkers of oat intake: a pharmacokinetic study of solid and liquid oat consumption under single and repeated dose conditions. Nutr J. 2025 Sep 9;24(1):136. doi: 10.1186/s12937-025-01204-7. PMID 40926245